CLINICAL TRIAL: NCT04733586
Title: Comparison Between Single Shot Ultrasonographic Guided Fascia Iliaca Block and Quadratus Lumborum Block in Hip Arthralgia. Comparative Double Blind Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mina Maher, Lecturer of anesthesia and ICU, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 122-1/2020
Record Dates: First submitted 2021-01-26; First posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fascia iliaca group (Active Comparator)
  Interventions: Procedure: Sonar guided fascia iliaca
- quadratus lumborum (Active Comparator)
  Interventions: Procedure: Sonar guided quadratus lumborum block

INTERVENTIONS:
Procedure: Sonar guided fascia iliaca — Sonar guided fascia iliaca
  Arms: fascia iliaca group
Procedure: Sonar guided quadratus lumborum block — Sonar guided quadratus lumborum block
  Arms: quadratus lumborum

SUMMARY:
hip arthralgia is a painful condition specially geriatric patients. Trail to alleviate pain using locoregional procedures

DETAILED DESCRIPTION:
hip arthralgia is a common presentation in many conditions as rheumatoid arthritis, systemic lupus . Pain is agonizing and disabling patinet to have normal life. we are considering fascial plane block versus quadratus lumborum block to dampen pain score.

ELIGIBILITY:
Inclusion Criteria:

* All candidates with hip arthalgia (primary or secondery)

Exclusion Criteria:

* History of warfarin or clopidogrel adminstration .
* patient on chemotherapy
* Cognitive disrder

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2021-02-20 (Estimated); Primary Completion 2021-05-20 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
pain score | one week and 3 months
  Visual analogue scale

IPD SHARING:
Plan to Share IPD: No